CLINICAL TRIAL: NCT02216266
Title: Monocenter, Double Blind, Randomised, Placebo Controlled Study to Evaluate Physostigmine for the Treatment of Delirium in Perioperative Intensive Care Medicine
Brief Title: Evaluation if Physostigmine Reduces Symptoms in Patients Who Has Developed a Delirium in Intensive Care After a Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PD Dr. Bertram Scheller (Other)
Collaborators: Goethe University (Other); Dr. Franz Köhler Chemie GmbH (study medication and labeling) (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr. Bertram Scheller, PD MD Bertram Scheller, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DELIcu; 2012-004082-41 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2014-08-13 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Suspected Delirium After Elective or Emergency Heart Surgery; CAM-ICU Diagnosed Delirium
Keywords: Delirium; CAM-ICU
MeSH Terms: conditions — Delirium | interventions — Physostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physostigmine (Active Comparator): Physostigmine administered intravenously at a dose of 24 mg + 25 min a 0,04 mg/kg milligram(s)/kilogram
  Interventions: Drug: Physostigmine
- Sodium Chloride solution (Placebo Comparator): solution administered intravenously 24 mg + 25 min a 0,04 mg/kg milligram(s)/kilogram
  Interventions: Other: Sodium Chloride solution

INTERVENTIONS:
Drug: Physostigmine
  Other Names: Anticholium
  Arms: Physostigmine
Other: Sodium Chloride solution
  Other Names: NaCl solution as Placebo comparator
  Arms: Sodium Chloride solution

SUMMARY:
Evaluation if physostigmine reduces symptoms in patients who has developed a delirium in Intensive care after a surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged > 18 years, < 85 years of ICU C1 after elective or emergency heart surgery with or without extracorporeal circulation (heart-lung machine and/or extracorporeal membrane oxygenation), with suspected delirium. (May be suspected if a patient does not show adequate improvement of vigilance 24 h after adequate reduction or stop of sedative medicine)
* Patients (>18a, <85a) with CAM-ICU diagnosed delirium
* Patients of legal capacity and patients with appointed representative

Exclusion Criteria:

* Asthma
* hypersensitivity against Physostigmine salicylate, Sodium metabisulfite, Nitrogen
* gangrene mechanical obstipation
* mechanical urinary retention
* Dystrophia myotonica
* Depolarization block after depolarising muscle relaxants
* Intoxications with "irreversibly acting" cholinesterase inhibitors
* closed head trauma
* obstructions at gastro-intestinal tract and at urinary tract
* neurological diseases
* left ventricular ejection fraction < 40%
* Simultaneous Participation in other clinical trials or participation ind other clinical trials in the last 30 days
* untreated coronary heart disease
* wish to have children, pregnancy or nursing
* patients with addictive disorder in medical history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of vigilance or symptoms of the delirium measured by Richmond Agitation Sedation Score (RASS) | baseline to 48 hours after administration

SECONDARY OUTCOMES:
reduction of weaning time at mechanical ventilator of patients with symptoms of delirium | baseline to 48 hours after administration
change in the spontaneous EEG and auditory evoked potentials | baseline to 48 hours after administration
  for the spontaneous EEG, we expect a shift in the frequency characteristics, measure is the spectrogram, more precisely the amplitude per frequency (band) and the phase information derived via Fourier Transform and Wavelet transformation
  The paradigm of the auditory stimulation is a roving paradigm (Science 13 May 2011:
  Vol. 332 no. 6031 pp. 858-862 DOI: 10.1126/science.1202043
  •Report Preserved Feedforward But Impaired Top-Down Processes in the Vegetative State Melanie Boly1,2,*, Marta Isabel Garrido2, Olivia Gosseries1, Marie-Aurélie Bruno1, Pierre Boveroux3, Caroline Schnakers1, Marcello Massimini4, Vladimir Litvak2, Steven Laureys1, Karl Friston2) Measures will be differences in the mismatch negativity and in the phase synchronization between electrodes
impact of the variability of heart rate | baseline to 48 hours
  heart rate variability is a dimensionless parameter, assessing the variability of the heart rate from ECG measures (Heart Rate Variability Conny M. A. van Ravenswaaij-Arts, MD; Louis A. A. Kollee, MD, PhD; Jeroen C. W. Hopman, MSc; Gerard B. A. Stoelinga, MD, PhD; and Herman P. van Geijn, MD, PhD [+-] Article and Author Information
  Ann Intern Med. 1993;118(6):436-447. doi:10.7326/0003-4819-118-6-199303150-00008 )
change in development of muscular force | baseline up to 48 hours
  muscular force is measured with a force gauge, measured in [Newton]
Occurence of Adverse events | baseline to 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Scheller, MD, Principal Investigator — Department of Anesthesiology, Intensive-Care Medicine and Pain Therapy of Goethe-University Frankfurt
Locations (1):
- Department of Anesthesiology, Intensive-Care Medicine and Pain Therapy, Frankfurt, Hessia, Germany